CLINICAL TRIAL: NCT07084376
Title: A Multicenter, Parallel-group, Randomized Controlled Trial to Assess the Efficacy of Two Different Educational Approaches on Intermittent Catheter-related Acceptance and Patient-Reported Outcome Measures (PROMs): RElax & feeL at EASE (RELEASE)
Brief Title: RElax & feeL at EASE (RELEASE)
Acronym: RELEASE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stefania Musco (Other)
Responsible Party: Sponsor-Investigator, Stefania Musco, MD, Careggi Hospital
Organization: Careggi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RELEASE
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Incontinence; Neurogenic Bladder Dysfunction; Urinary Retention
Keywords: Intermittent catheterization; Self-catheterization; Patient education; Adherence; Acceptance; Male urology
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: This is a multicenter, parallel-group, randomized controlled trial with two arms. Participants are randomized 1:1 to either an enhanced educational intervention group (informational booklet, video, and standard training) or a control group receiving standard training only. The parallel design allows for direct comparison of outcomes between these two educational strategies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Educational Program for Intermittent Catheterization (Experimental): Participants in this arm will receive an enhanced educational intervention comprising an informational booklet, a video tutorial specifically designed for self-managed intermittent catheterization (IC), and standard clinical practice training. This comprehensive approach aims to improve psychological acceptance, adherence, and self-efficacy in performing IC
  Interventions: Other: Enhanced Educational Program for Intermittent Catheterization
- Standard Education Group (Active Comparator): Participants receive standard clinical practice training for self-managed intermittent catheterization (IC) as typically provided in routine care settings. This arm serves as the active comparator to evaluate the additional impact of the enhanced educational intervention.
  Interventions: Other: Standard Education Group

INTERVENTIONS:
Other: Enhanced Educational Program for Intermittent Catheterization — Participants in this group receive an enhanced educational program for intermittent catheterization (IC), including an informational booklet, a specifically designed video tutorial, and standard clinical practice training. The program aims to improve psychological acceptance, adherence, and self-efficacy by providing comprehensive and patient-centered educational materials in addition to standard care.
  Arms: Enhanced Educational Program for Intermittent Catheterization
Other: Standard Education Group — Participants in this group will receive standard clinical practice training for intermittent catheterization (IC), as routinely provided in participating healthcare centers. This training focuses on basic procedural skills and practical education necessary to perform IC independently, without additional enhanced educational materials such as booklets or video tutorials.
  Arms: Standard Education Group

SUMMARY:
This multicenter, parallel-group, randomized controlled trial (RELEASE) aims to evaluate the efficacy of two educational approaches on acceptance and adherence to intermittent catheterization (IC) among adult male patients. Participants requiring IC training will be randomized to either an enhanced educational intervention (informational booklet, video tutorial, and standard training) or standard clinical practice training alone. The primary outcome is the change in Intermittent Catheterization Acceptance Test (I-CAT) scores over three months. Secondary outcomes include adherence (I-CAS), urinary symptoms (USQNB-IC), patient autonomy, satisfaction with assistive technology (QUEST), and functional abilities. The study seeks to identify the most effective educational strategy to improve psychological acceptance, promote adherence, and reduce complications in patients performing IC, ultimately supporting patient-centered care and health system efficiency.

DETAILED DESCRIPTION:
This multicenter, randomized controlled trial (RELEASE study) investigates the effectiveness of two different educational approaches to improve acceptance and adherence to intermittent catheterization (IC) among adult male patients who require IC training. Participants will be randomly assigned to one of two groups: an intervention group receiving an enhanced educational program (including an informational booklet, video tutorial, and standard clinical training) and a control group receiving only standard clinical practice training.

The study will enroll adult male patients with an indication for self-managed intermittent catheterization and who are physically and cognitively able to learn IC techniques. The primary outcome measure is the change in Intermittent Catheterization Acceptance Test (I-CAT) scores at three months (T2) compared to baseline (T0).

Secondary outcomes include adherence measured using the Intermittent Catheterization Adherence Scale (I-CAS), urinary symptoms evaluated with the USQNB-IC, patient autonomy, satisfaction with assistive technology (QUEST 2.0), and overall functional abilities. Additional data such as socio-demographic characteristics and medical history will also be collected.

The trial seeks to provide evidence on the most effective educational strategy to support psychological acceptance and sustained adherence to IC, reduce complications, and promote greater patient autonomy. By addressing educational gaps, the study aims to enhance patient-centered care and optimize resource use within the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years or older.
* Diagnosed with neurogenic bladder requiring self-managed intermittent catheterization (IC).
* Currently performing IC or newly prescribed IC.
* Able to provide informed consent and understand study instructions.
* Able to understand and complete study questionnaires in Italian.

Exclusion Criteria:

* Presence of cognitive impairment limiting ability to understand or perform IC independently.
* Severe upper limb motor deficits preventing independent catheterization.
* Active urinary tract infection at baseline.
* Participation in another interventional study that could interfere with outcomes.
* Any condition that, in the opinion of the investigators, makes the patient unsuitable for study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who identify as male and correspond to the biological sex assigned at birth (male) are eligible to participate in this study.
Enrollment: 64 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Intermittent Catheterization Acceptance (I-CAT) Score | Baseline (T0) to 3 months (T2)
  Change in psychological acceptance of intermittent catheterization measured using the Intermittent Catheterization Acceptance Test (I-CAT). The I-CAT assesses acceptance attitudes toward IC, including psychological readiness and emotional adaptation. Higher scores indicate greater acceptance.

SECONDARY OUTCOMES:
Adherence to Intermittent Catheterization (I-CAS Score) | Baseline (T0) to 3 months (T2)
  Adherence to intermittent catheterization practices measured by the Intermittent Catheterization Adherence Scale (I-CAS). The scale evaluates the frequency and consistency of IC behaviors. Higher scores indicate greater adherence.
Urinary Symptoms Severity (USQNB-IC) | Baseline (T0) to 3 months (T2)
  Severity of urinary symptoms measured by the Urinary Symptom Questionnaire for Neurogenic Bladder-Intermittent Catheterization (USQNB-IC). This assesses frequency and severity of symptoms related to bladder dysfunction and catheterization.
Patient Autonomy Level | Baseline (T0) to 3 months (T2)
  Self-reported autonomy in performing intermittent catheterization, assessed through specific questions evaluating confidence and independence in IC management.
Satisfaction with Assistive Technology (QUEST 2.0) | 3 months (T2)
  Satisfaction with assistive technology measured using the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0). Higher scores reflect greater satisfaction with IC-related aids and support tools.
Overall Functional Abilities | Baseline (T0) to 3 months (T2)
  Changes in overall functional abilities assessed through patient self-reports on mobility, self-care, and daily activities impacted by IC.

IPD SHARING:
Plan to Share IPD: No
Given the nature of your intervention (behavioral educational intervention on intermittent catheterization) and local privacy considerations, individual participant data (IPD) will not be shared publicly.

REFERENCES:
- [Background] Vecchio M, Chiaramonte R, DI Benedetto P. Management of bladder dysfunction in multiple sclerosis: a systematic review and meta-analysis of studies regarding bladder rehabilitation. Eur J Phys Rehabil Med. 2022 Jun;58(3):387-396. doi: 10.23736/S1973-9087.22.07217-3. Epub 2022 Feb 1. PMID 35102733
- [Background] van der Woude DR, Ruyten T, Bartels B. Reliability of Muscle Strength and Muscle Power Assessments Using Isokinetic Dynamometry in Neuromuscular Diseases: A Systematic Review. Phys Ther. 2022 Oct 6;102(10):pzac099. doi: 10.1093/ptj/pzac099. PMID 35899532
- [Background] Tractenberg RE, Groah SL, Rounds AK, Ljungberg IH, Schladen MM. Preliminary validation of a Urinary Symptom Questionnaire for individuals with Neuropathic Bladder using Intermittent Catheterization (USQNB-IC): A patient-centered patient reported outcome. PLoS One. 2018 Jul 10;13(7):e0197568. doi: 10.1371/journal.pone.0197568. eCollection 2018. PMID 29990375
- [Background] Tornic J, Panicker JN. The Management of Lower Urinary Tract Dysfunction in Multiple Sclerosis. Curr Neurol Neurosci Rep. 2018 Jun 28;18(8):54. doi: 10.1007/s11910-018-0857-z. PMID 29956001
- [Background] Sutton G, Shah S, Hill V. Clean intermittent self-catheterisation for quadriplegic patients--a five year follow-up. Paraplegia. 1991 Oct;29(8):542-9. doi: 10.1038/sc.1991.78. PMID 1775361
- [Background] Reuben DB, Magasi S, McCreath HE, Bohannon RW, Wang YC, Bubela DJ, Rymer WZ, Beaumont J, Rine RM, Lai JS, Gershon RC. Motor assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S65-75. doi: 10.1212/WNL.0b013e3182872e01. PMID 23479547
- [Background] Milligan J, Goetz LL, Kennelly MJ. A Primary Care Provider's Guide to Management of Neurogenic Lower Urinary Tract Dysfunction and Urinary Tract Infection After Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2020 Spring;26(2):108-115. doi: 10.46292/sci2602-108. PMID 32760189
- [Background] Manack A, Motsko SP, Haag-Molkenteller C, Dmochowski RR, Goehring EL Jr, Nguyen-Khoa BA, Jones JK. Epidemiology and healthcare utilization of neurogenic bladder patients in a US claims database. Neurourol Urodyn. 2011 Mar;30(3):395-401. doi: 10.1002/nau.21003. Epub 2010 Sep 29. PMID 20882676
- [Background] Lapides J, Diokno AC, Lowe BS, Kalish MD. Followup on unsterile intermittent self-catheterization. J Urol. 1974 Feb;111(2):184-7. doi: 10.1016/s0022-5347(17)59922-x. No abstract available. PMID 4810761
- [Background] Guinet-Lacoste A, Charlanes A, Chesnel C, Blouet E, Tan E, Le Breton F, Amarenco G. Intermittent Catheterization Adherence Scale (ICAS): A new tool for the evaluation of patient adherence with clean intermittent self-catheterization. Neurourol Urodyn. 2018 Nov;37(8):2753-2757. doi: 10.1002/nau.23746. Epub 2018 Jun 28. PMID 29953666
- [Background] Fitzpatrick MA, Solanki P, Wirth M, Weaver FM, Suda KJ, Burns SP, Safdar N, Collins E, Evans CT. Perceptions, experiences, and beliefs regarding urinary tract infections in patients with neurogenic bladder: A qualitative study. PLoS One. 2023 Nov 1;18(11):e0293743. doi: 10.1371/journal.pone.0293743. eCollection 2023. PMID 37910578
- [Background] Fitzpatrick MA, Solanki P, Wirth M, Weaver FM, Suda KJ, Burns SP, Safdar N, Collins E, Evans CT. Knowledge, perceptions, and beliefs about urinary tract infections in persons with neurogenic bladder and impacts on interventions to promote person-centered care. Spinal Cord. 2024 May;62(5):221-227. doi: 10.1038/s41393-024-00972-z. Epub 2024 Mar 7. PMID 38454065
- [Background] Blanc BF, Rodriguez-Almagro J, Lorenzo-Garcia C, Alcaraz-Zomeno E, Fernandez-Llorente G, Baixauli-Puig M, Martin-Bermejo MV, Estudillo-Gonzalez F, Ortega-Checa MA, Lluesma-Martinez V, Ferrandez-Franco G, Benito-Santos B, Rodriguez-Diaz M, Torres-Bacete A, Guerrero-Andrades MC, Louis-Lauture MP, Jimenez-Mayorga I, Serrano-Abielar R, Garrido-Mora MA, Barcia-Barrera F, Asensio-Malo G, Morcillo-Marin M, Tendero-Ruiz S, Hernandez-Martinez A. Quality of Life and Autonomy in Patients with Intermittent Bladder Catheterization Trained by Specialized Nurses. J Clin Med. 2021 Aug 30;10(17):3909. doi: 10.3390/jcm10173909. PMID 34501357
- [Background] Berardi A, Marquez MA, Ottone L, Ruotolo I, Panuccio F, Tofani M, Gonzalez-Bernal J, Galeoto G. Italian translation, cultural adaptation, and validation of the Intermittent Catheterization Acceptance Test (I-CAT). Clin Ter. 2023 Jan-Feb;174(1):8-13. doi: 10.7417/CT.2023.5002. PMID 36655638